CLINICAL TRIAL: NCT00334841
Title: Leptin and Cytokines in Diabetic Pregnancy - Physiologic or Pathogenic Role
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 0507874356- HMO-CTIL
Record Dates: First submitted 2006-06-05; First posted 2006-06-08 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2006-05

CONDITIONS: Gestational Diabetes Mellitus; Preeclampsia; Placental Hypoxia
MeSH Terms: conditions — Diabetes, Gestational; Pre-Eclampsia

SUMMARY:
Leptin, a circulating hormone expressed abundantly in adipose tissue, has been reported to be a satiety factor. In addition, it has been shown to increase during pregnancy in maternal blood, parallel to increase in body fat mass, to correlate with fetal body weight gain and to fall down to basal levels after delivery.

Little is known about leptin levels in pregnant women with preexisting or gestational diabetes and their relationship with fetal and postnatal growth and perinatal complications.

Therefore, the proposed study aims to understand and characterize the role of leptin in gestational diabetes mellitus as well as the relationship between leptin, cytokines and the pathophysiological complications during diabetic pregnancy. Specifically, we will evaluate 60 pregnant women both in Germany and in Israel and evaluate serum levels and mRNA of leptin, cytokines (inflammatory as well as Th1 and Th2) and correlate them to maternal changes of body weight and birth weight in women of various degrees of glucose tolerance and with various degrees of metabolic control during pregnancy; relationship between serum and umbilical cord vein concentrations of leptin, cytokines and metabolic variables; placental expression of leptin, leptin receptor, selected cytokines, GLUT1 and 4 and relationship to leptin in serum and umbilical cord plasma; comparison between all above parameters of German and Israeli pregnant women.

The results of this new and systematic study will shed light on the role of leptin and cytokines in the development of glucose disturbances during pregnancy and the perinatal outcome of women with gestational or preexisting diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

random glucose challenge test (GCT): 50 g of glucose are orally given at any time of the day. The results are considered as positive if the capillary blood glucose concentrations 1 hour after the load are >130 mg/dl. Those with normal results serve as control group

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Elchalal, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Lappas M, Yee K, Permezel M, Rice GE. Release and regulation of leptin, resistin and adiponectin from human placenta, fetal membranes, and maternal adipose tissue and skeletal muscle from normal and gestational diabetes mellitus-complicated pregnancies. J Endocrinol. 2005 Sep;186(3):457-65. doi: 10.1677/joe.1.06227. PMID 16135665